CLINICAL TRIAL: NCT06632327
Title: Perioperative Versus Adjuvant Systemic Therapy in Patients With Resectable Non-Small Cell Lung Cancer - PROSPECT LUNG
Brief Title: Comparing Impact of Treatment Before or After Surgery in Patients With Stage II-IIIB Resectable Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTIU2317-A082304-S2402; NCI-2024-06356 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Resectable Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative; Cisplatin; Carboplatin; Pemetrexed; Gemcitabine; Docetaxel; Vinorelbine; Nivolumab; pembrolizumab; atezolizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (surgery, adjuvant therapy) (Experimental): SURGERY: Patients undergo surgery within 28 days of registration.
  ADJUVANT THERAPY: Patients receive platinum-based doublet chemotherapy (cisplatin, carboplatin, pemetrexed, gemcitabine, docetaxel, and/or vinorelbine) for up to 4 cycles and immune checkpoint inhibitor therapy (nivolumab, pembrolizumab, and/or atezolizumab) for up to 1 year in the absence of disease progression or unacceptable toxicity according to current approved guidelines.
  Patients also undergo CT throughout the study and may undergo MRI and/or PET/CT at screening.
  Interventions: Procedure: Surgical Procedure; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Docetaxel; Drug: Vinorelbine; Drug: Nivolumab; Drug: Pembrolizumab; Drug: Atezolizumab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Arm 2 (neoadjuvant therapy, surgery, adjuvant therapy) (Experimental): NEOADJUVANT THERAPY: Within 28 days of registration, patients receive platinum-based doublet chemotherapy (cisplatin, carboplatin, pemetrexed, gemcitabine, docetaxel, and/or vinorelbine) for up to 4 cycles in combination with immune checkpoint inhibitor (nivolumab, pembrolizumab, and/or atezolizumab) according to current approved guidelines.
  SURGERY: Patients undergo surgery.
  ADJUVANT THERAPY: Patients receive immune checkpoint inhibitor therapy (nivolumab, pembrolizumab, and/or atezolizumab) for up to 1 year in the absence of disease progression or unacceptable toxicity according to current approved guidelines.
  Patients also undergo CT throughout the study and may undergo MRI and/or PET/CT at screening.
  Interventions: Procedure: Surgical Procedure; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Docetaxel; Drug: Vinorelbine; Drug: Nivolumab; Drug: Pembrolizumab; Drug: Atezolizumab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Surgical Procedure — undergo surgery
Drug: Cisplatin — Give cisplatin
Drug: Carboplatin — Give Carboplatin
Drug: Pemetrexed — Give Pemetrexed
Drug: Gemcitabine — Give Gemcitabine
Drug: Docetaxel — Give Docetaxel
Drug: Vinorelbine — Give Vinorelbine
Drug: Nivolumab — Give Nivolumab
Drug: Pembrolizumab — Give Pembrolizumab
Drug: Atezolizumab — Give Atezolizumab
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CT Scan; CAT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: PET Scan

SUMMARY:
This phase III trial compares standard therapy given after surgery (adjuvant) to standard therapy given before and after surgery (perioperative) in treating patients with stage II-IIIB non-small cell lung cancer (NSCLC) that can be removed by surgery (resectable). The usual approach for patients with resectable NSCLC is chemotherapy and/or immunotherapy before surgery, after surgery, or both before and after surgery. This study is being done to find out which approach is better at treating patients with lung cancer. Treatment will be administered according to the current standard of care at the time of enrollment. Chemotherapy options may include cisplatin, carboplatin, pemetrexed, gemcitabine, docetaxel, and vinorelbine at standard doses according to the treating physician. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Pemetrexed is in a class of medications called antifolate antineoplastic agents. It works by stopping cells from using folic acid to make deoxyribonucleic acid (DNA) and may kill tumor cells. Gemcitabine is a chemotherapy drug that blocks the cells from making DNA and may kill tumor cells. Docetaxel is in a class of medications called taxanes. It stops tumor cells from growing and dividing and may kill them. Other chemotherapy drugs, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading . Immunotherapy with monoclonal antibodies, such as nivolumab, pembrolizumab, and atezolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Starting treatment with chemotherapy and immunotherapy prior to surgery and continuing treatment after surgery may be a more effective treatment option than adjuvant therapy alone in patients with stage II-IIIB resectable NSCLC.

DETAILED DESCRIPTION:
The primary and secondary objectives of the study:

PRIMARY OBJECTIVE:

I. To compare the 3-year real-world event-free survival (rwEFS) rate and overall survival (OS) between perioperative and adjuvant immunotherapy-based treatment for patients with resectable non-small cell lung cancer (dual endpoints).

SECONDARY OBJECTIVES:

I. To compare the rates of surgical resection between the two arms. II. To compare the rates of complete resection (R0) between the two arms. III. To summarize and compare rates of adverse events (AEs) resulting in permanent treatment discontinuation, hospitalization, or death between the two arms.

IV. To evaluate the association between locally defined pathological complete response (pCR) and rwEFS in patients randomized to the perioperative arm (arm 2).

V. To compare the rwEFS post 3-years from randomization between the two arms among patients who do not experience an event by 3 years.

EXPLORATORY OBJECTIVES:

I. To compare outcomes according to the systemic therapy administered on each arm.

II. To compare the sites of relapse between the two treatment arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1:

SURGERY: Patients undergo surgery within 28 days of registration.

ADJUVANT THERAPY: Patients receive platinum-based doublet chemotherapy (cisplatin, carboplatin, pemetrexed, gemcitabine, docetaxel, and/or vinorelbine) for up to 4 cycles and immune checkpoint inhibitor therapy (nivolumab, pembrolizumab, and/or atezolizumab) for up to 1 year in the absence of disease progression or unacceptable toxicity according to current approved guidelines.

ARM 2:

NEOADJUVANT THERAPY: Within 28 days of registration, patients receive platinum-based doublet chemotherapy (cisplatin, carboplatin, pemetrexed, gemcitabine, docetaxel, and/or vinorelbine) for up to 4 cycles in combination with immune checkpoint inhibitor (nivolumab, pembrolizumab, and/or atezolizumab) according to current approved guidelines.

SURGERY: Patients undergo surgery.

ADJUVANT THERAPY: Patients receive immune checkpoint inhibitor therapy (nivolumab, pembrolizumab, and/or atezolizumab) for up to 1 year in the absence of disease progression or unacceptable toxicity according to current approved guidelines.

Patients also undergo computed tomography (CT) throughout the study and may undergo magnetic resonance imaging (MRI) and/or positron emission tomography (PET)/CT at screening.

After completion of study treatment, patients are followed up every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed surgically resectable stage IIA to IIIB NSCLC according to the American Joint Committee on Cancer (AJCC) 9th edition (stage IIA to IIIB NSCLC up to single station N2, according to the AJCC 8th edition)

  * Note: Patients with resectable stage N2a or T4 are eligible, but patients with stage N2b or N3 are not eligible. Patients with known EGFR or ALK alterations are excluded
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (or Karnofsky ≥ 60%)
* No prior systemic treatment for NSCLC within 5 years except stage 1 and 2 cancers treated with curative intent
* No treatment for another malignancy within 3 years prior to registration, except for stage 1 or 2 cancers treated for curative intent; patients must be disease free for one year prior to registration. Patients with non-melanoma skin cancer, urothelial carcinoma in situ (Tis), noninvasive papillary carcinoma of the urinary bladder (Ta), prostatic intraepithelial neoplasia (PIN), ductal carcinoma in situ (DCIS) of the breast, or cervical intraepithelial neoplasia (CIN) of the uterine cervix are also eligible
* No active autoimmune disease, interstitial lung disease, or transplant that precludes safe treatment with immune checkpoint inhibitors
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
3-year real-world event-free survival (rwEFS) | From the date of randomization to the date of the first of the following events: failure to undergo resection for any reason, recurrence or progression at any time after surgery, or death from any cause, assessed at 3 years
  Time to event analyses will be summarized using the Kaplan-Meier method, where both the stratified and unstratified log-rank test will be used to compare the distributions across the treatment arms. For the primary analysis of 3-year rwEFS rate, we will compare the rwEFS curves at 3 years, using the difference in Kaplan-Meier estimates for the survival functions. The test statistic will be derived from the difference in the estimated Kaplan-Meier values between two arms at 3 years, using the Greenwood estimate of the variances. rwEFS rates at 1 year, 2 years, and 5 years will also be reported, along with 95% confidence intervals. The comparison of the rwEFS post 3-years between the two arms among patients who do not experience an event by 3 years, will involve assessing the probability of a longer rwEFS on the perioperative arm. Non-parametric estimation and inference methods will be used for analysis.
Overall survival (OS) | From randomization until death from any cause, assessed up to 10 years
  Time to event analyses will be summarized using the Kaplan-Meier method, where both the stratified and unstratified log-rank test will be used to compare the distributions across the treatment arms. OS rates at 1 year, 2 years, and 5 years will also be reported, along with 95% confidence intervals.

SECONDARY OUTCOMES:
Rates of surgical resection | Up to 10 years.
  Rates of resection will be tabulated and compared between the arms using chi-square tests or Fisher's exact tests. Univariable Cox models stratified by the stratification factors used in the randomization will be used to understand the impact of baseline covariates, resection status and systemic treatments on outcomes.
Rates of complete resection (R0) | Up to 10 years.
  Rates of R0 resection will be tabulated and compared between the arms using chi-square tests or Fisher's exact tests. Univariable Cox models stratified by the stratification factors used in the randomization will be used to understand the impact of baseline covariates, resection status and systemic treatments on outcomes.
Incidence of adverse events (AEs) | Up to 10 years.
  Adverse events will be recorded using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 for each patient. Frequency tables and summary statistics will be used to determine the overall patterns within and across the arms.
Pathological complete response (pCR) | Up to 10 years
  Pathologic complete response is defined as having no viable invasive cancer in the lung and lymph nodes (ypT0 ypN0 or ypT0/is ypN0) based on guidelines published by National Comprehensive Cancer Network and International Association for the Study of Lung Cancer. Cox regression models will be used to evaluate the association between pCR and rwEFS in perioperative arm (arm 2). The hazard ratio and corresponding 95% confidence interval will be reported. Multivariable landmark and time dependent models will be subsequently explored.

OTHER OUTCOMES:
Estimates of treatment effect by sex | Up to 10 years.
  Estimates of 3-year rwEFS rates and hazard ratio for OS and the corresponding 95% confidence intervals (CIs) will be evaluated by sex.
Estimates of treatment effect by race | Up to 10 years
  Estimates of 3-year rwEFS rates and hazard ratio for OS and the corresponding 95% confidence intervals (CIs) will be evaluated by race.
Estimates of treatment effect by ethnicity | Up to 10 years
  Estimates of 3-year rwEFS rates and hazard ratio for OS and the corresponding 95% confidence intervals (CIs) will be evaluated by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, MD, Study Chair — Alliance for Clinical Trials in Oncology; Raid Aljumaily, MD, Study Chair — Alliance for Clinical Trials in Oncology; Linda Martin, MD, Study Chair — Alliance for Clinical Trials in Oncology
Locations (369):
- United States (369):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Enloe Medical Center, Chico, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Orlando Health Cancer Institute - Lake Mary, Lake Mary, Florida
  - The Watson Clinic, Lakeland, Florida
  - Health Central, Ocoee, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Reid Health, Richmond, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Tufts Medical Center Cancer Center Stoneham, Stoneham, Massachusetts
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Veteran's Affairs Medical Center - Saint Louis, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Benefis Helena Specialty Center, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Glens Falls Hospital, Glens Falls, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Saint Michael Cancer Center, Silverdale, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Memorial Hospital of Laramie County, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming